CLINICAL TRIAL: NCT06684795
Title: An Open-label, Non-randomized, Single Dose, Phase II Trial of FG001 (an Optical Imaging Agent) for Localization of Meningiomas or Presumed Low-Grade Gliomas Scheduled for Neurosurgery
Brief Title: FG001 in Subjects with Meningiomas or Presumed Low-Grade Gliomas Scheduled for Neurosurgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jane Skjøth-Rasmussen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RH-FG001-001
Record Dates: First submitted 2024-06-20; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-06

CONDITIONS: Low-grade Glioma; Meningioma; Glioma
MeSH Terms: conditions — Meningioma; Glioma

STUDY DESIGN:
Intervention Model Description: A total of 40 patients are planned for enrolment. The study will include two arms, where one arm will consist of patients with presumed low-grade gliomas (pLGG) and one with meningiomas.
  Initially, 20 patients (pLGG=10 and meningioma=10) will be enrolled in the trial followed by an interim analysis. Here, further modifications in the trial with respect to dose administration time and administered dose is possible before enrolment of the last 20 patients (pLGG=10 and meningioma=10).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Presumed low-grade glioma (Experimental)
  Interventions: Drug: FG001 prior to surgery
- Meningioma (Experimental)
  Interventions: Drug: FG001 prior to surgery

INTERVENTIONS:
Drug: FG001 prior to surgery — Patients will receive a single intravenous injection of 36 mg FG001 administered the day before surgery.

SUMMARY:
In neurosurgery both the diffusely infiltrated gliomas of the brain as well as the border towards healthy tissue in the meninges is a challenge. For the high-grade contrast enhanced gliomas fluorescent drugs like Gliolan have been used in several years and proved its clinical value. For non-contrast enhanced gliomas, like low-grade glioma, no such drug exist. The transition zone towards healthy non-tumor cell infiltrated brain in such low-grade gliomas is extremely difficult but for these patients their prognosis depends on the amount of non-healthy tissue left behind. Also, in benign tumors as meningioma the complete resection including infiltrated meninges is of importance for the cure of the disease. None of the existing fluorescent drug is useful or approved for these tumors.. Hence a medicinal product that will fulfil the criteria for a safe and reliable fluorescent drug to guide the surgery to the boundaries of the infiltration with tumor cells is highly warranted.

DETAILED DESCRIPTION:
The drug FG001 (ICG-Glu-Glu-AE105), a uPAR-targeting fluorescent drug, has been tested in patients with high-grade glioma as part of a First-in-human clinical trial and demonstrated an excellent safety profile and efficacy results. Animal studies have indicated uptake of FG001 in low-grade glioma while uptake has been shown in one clinical case of meningioma providing the basis for this trial.

Consequently, the investigators intend to test the ability of FG001 to reliably fluoresce in patients with presumed low-grade glioma or meningioma.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be entered into this trial only if they meet all the following criteria:

1. Subjects diagnosed with primary brain tumor on MRI suggestive of, meningioma or presumed low-grade glioma (pLGG)*
2. Scheduled for neurosurgery with the objective to remove cancer tissue
3. Subjects aged 18 years or older
4. Capable of understanding and giving written informed consent
5. Women of childbearing potential must agree to use an adequate method of contraception during the trial and for 30 days after the end-of-trial visit. Adequate methods of contraception include intrauterine device or hormonal contraception (oral contraceptive pill, depot injections or implant, transdermal depot patch or vaginal ring). To be considered sterilised or infertile, females must have undergone surgical sterilisation (bilateral tubectomy, hysterectomy or bilateral ovariectomy) or be post-menopausal (defined as at least 12 months amenorrhoea; may be confirmed with follicle-stimulating hormone [FSH] test if there is doubt)
6. Male subjects must commit to use barrier contraception (e.g., condom) during the trial and for 30 days after the end-of-trial visit.
7. Subject must not previously have received the trial drug (FG001)
8. Subjects must have normal organ and bone marrow function and be appropriate surgical candidates per site standard of care (SOC) *Presumed low-grade gliomas in this protocol are defined as diffusely infiltrated non-contrast enhancing tumors on MRI. Patients with known LGG scheduled for re-surgery or primary surgery after a diagnostic biopsy may also be included.

Exclusion Criteria:

1. Any known allergy or hypersensitivity to indocyanine green (ICG)
2. Female subjects who are pregnant or breast-feeding (pregnancy test positive prior to inclusion (or if breast-feeding willing to pause breast feeding during trial and for 30 days
3. Overall performance status or co-morbidity deeming the subject unfitted for participation in the trial as judged by the Investigator
4. Pre-existing hepatic and/or renal insufficiency

   * INR above 1.7
   * Estimated GFR (eGFR) below 45 ml/min/1.73m2
5. Unwilling or unable to follow the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary objective | 24 months
  The primary objective is to evaluate the sensitivity of FG001 for detection of tumor tissue from meningioma and pLGG. The sensitivity will be evaluated as the proportion of subjects with fluorescent tumors given the tumor has been histologically verified.

SECONDARY OUTCOMES:
Secondary outcome | 24 months
  The efficacy of FG001 as a tumor imaging agent and safety will be monitored. The efficacy is examined by the sensitivity and specificity. Sensitivity is defined as the probability that a test result is positive when the subject has the disease, while specificity is the probability that a test result is negative when the patient does not have the disease. Safety is determined by physical examinations, laboratory samples and the incidence and severity of the Adverse events (AEs), which are evaluated by National Cancer Institute (NCI) Common Technology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Skjøth-Rasmussen, MD, PhD, Principal Investigator — Department of neurosurgery, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Witt Hamer PC, Robles SG, Zwinderman AH, Duffau H, Berger MS. Impact of intraoperative stimulation brain mapping on glioma surgery outcome: a meta-analysis. J Clin Oncol. 2012 Jul 10;30(20):2559-65. doi: 10.1200/JCO.2011.38.4818. Epub 2012 Apr 23. PMID 22529254
- [Background] Skjoth-Rasmussen J, Azam A, Larsen CC, Scheie D, Juhl K, Kjaer A. A new uPAR-targeting fluorescent probe for optical guided intracranial surgery in resection of a meningioma-a case report. Acta Neurochir (Wien). 2022 Jan;164(1):267-271. doi: 10.1007/s00701-021-05051-3. Epub 2021 Nov 8. PMID 34748074
- [Background] Skjøth-Rasmussen J, Azam A, Juhl K, Ginsborg S, Kryspin Sørensen M, Sølling C, Larsen CC, Scheie D, Kjaer A. First-in-human study of a novel Upar-targeted imaging agent (FGO01) for visualization of malignant glioma during surgery. Brain and Spine. 2022.